CLINICAL TRIAL: NCT06124859
Title: Assessment of Exercise Tolerance and Lower-limb Muscle Power in Patients With Chronic Respiratory Disease: a Multicenter Validity Study
Brief Title: Exercise Tolerance and Lower-limb Muscle Power in Patients With Chronic Respiratory Disease
Acronym: VTEP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Lille Catholic University (Other)
Collaborators: University of Lille Nord de France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC-P00120
Record Dates: First submitted 2023-10-30; First posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Pulmonary Fibrosis; Pulmonary Disease, Chronic Obstructive
Keywords: Six minutes stepper test (6MST); 5-times sit to stand test (5STS); Chronic obstructive pulmonary disease (COPD); Pulmonary Fibrosis
MeSH Terms: conditions — Pulmonary Fibrosis; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with a diagnosis of COPD (GOLD II- V) or pulmonary fibrosis (>6 months). (Experimental)
  Interventions: Other: Functional capacity tests

INTERVENTIONS:
Other: Functional capacity tests — Maximal effort test on cycloergometer (1st visit)
  Maximal effort test, 6-minute stepper test, 6-minute walk test, 5-times sit to stand test. A minimum rest period of 15 minutes must be observed between these tests (2nd Visit)

SUMMARY:
The aim of this study is to validate the six minute Stepper Test (6MST) and the 5-repetition chair lift test (5STS) as measures of exercise tolerance and muscle power, respectively, in patients with chronic respiratory disease.

As the reproducibility of the tests has been studied and validated in previous studies, the objective is to investigate the validity of the 6MST and 5STS in comparison with their respective gold standards.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 and over
* With a diagnosis of chronic obstructive pulmonary disease (GOLD II - IV) or pulmonary fibrosis (>6 months).
* Able to understand and follow verbal instructions during tests
* Affiliated with a social security scheme
* Willing to participate in the study

Exclusion Criteria:

* Have a neurological, cardiovascular or balance disorder that could impair test performance.
* Having undergone respiratory rehabilitation within the last year.
* With unstable disease (recent exacerbation < 4 weeks).
* Pregnant and/or breast-feeding women
* Patients under guardianship or curatorship

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Oxygen consumption | 19 days
  Oxygen consumption will be measured using the Cortex Metamax 3B (MM3B) automated gas analysis system. Maximum oxygen consumption obtained at the end of six minutes step test (6MST) and compared with the maximum oxygen consumption obtained in the maximum cardiorespiratory exercise test performed on a cycloergometer (gold standard for measuring exercise tolerance). The 6MST aims at measuring the number of steps performed on a stepper in 6 minutes. A step is defined as a single complete movement of raising one foot and putting it down. The stepper is placed on the ground facing a wall to allow patients to maintain their balance by placing their fingers on the wall. The step height is set at 20 cm. Before starting the test, patients get accustomed to the stepper for 2 minutes. The protocol include a 3-minute rest period and a 6-minute stepping period.
Lower limb muscle power after Five Times Sit to Stand Test (5STS,) calculated by the ratio between STS mean velocity and STS mean force | 19 days
  The 5XSTS scoring is based on the amount of time (to the nearest decimal in seconds) a patient is able to transfer from a seated to a standing position and back to sitting five times. The lower the time to complete the test the better the outcome of the test.The Lower limb muscle power will be calculated by the ratio between STS mean velocity and STS mean force according to the following equation :
  Power 5STS = body mass x 0,9 x g x (Height x 0,5 - chair height)/(time 5STS x 0,1)
  *g = 9,81 m/s, body mass in kg et Height in meters.

SECONDARY OUTCOMES:
Heart rate after 6MST | 19 days
  The 6MST aims at measuring the number of steps performed on a stepper in 6 minutes. A step is defined as a single complete movement of raising one foot and putting it down. The stepper is placed on the ground facing a wall to allow patients to maintain their balance by placing their fingers on the wall. The step height is set at 20 cm. Before starting the test, patients get accustomed to the stepper for 2 minutes. The protocol include a 3-minute rest period and a 6-minute stepping period.This measurement will be compared with those measured during a 6-minute walk test (gold standard for field tests) and a maximal cardiorespiratory exercise test on a cycloergometer (gold standard for laboratory tests)
Oxygen saturation after 6MST | 19 days
  Oxygen saturation will be measured using the Cortex Metamax 3B (MM3B) automated gas analysis system. The 6MST aims at measuring the number of steps performed on a stepper in 6 minutes. A step is defined as a single complete movement of raising one foot and putting it down. The stepper is placed on the ground facing a wall to allow patients to maintain their balance by placing their fingers on the wall. The step height is set at 20 cm. Before starting the test, patients get accustomed to the stepper for 2 minutes. The protocol include a 3-minute rest period and a 6-minute stepping period.This measurement will be compared with those measured during a 6-minute walk test (gold standard for field tests) and a maximal cardiorespiratory exercise test on a cycloergometer (gold standard for laboratory tests)
Minute ventilation after 6MST | 19 days
  Minute ventilation will be measured using the Cortex Metamax 3B (MM3B) automated gas analysis system. The 6MST aims at measuring the number of steps performed on a stepper in 6 minutes. A step is defined as a single complete movement of raising one foot and putting it down. The stepper is placed on the ground facing a wall to allow patients to maintain their balance by placing their fingers on the wall. The step height is set at 20 cm. Before starting the test, patients get accustomed to the stepper for 2 minutes. The protocol include a 3-minute rest period and a 6-minute stepping period.This measurement will be compared with those measured during a 6-minute walk test (gold standard for field tests) and a maximal cardiorespiratory exercise test on a cycloergometer (gold standard for laboratory tests)
Respiratory rate after 6MST | 19 days
  Respiratory rate will be measured using the Cortex Metamax 3B (MM3B) automated gas analysis system. The 6MST aims at measuring the number of steps performed on a stepper in 6 minutes. A step is defined as a single complete movement of raising one foot and putting it down. The stepper is placed on the ground facing a wall to allow patients to maintain their balance by placing their fingers on the wall. The step height is set at 20 cm. Before starting the test, patients get accustomed to the stepper for 2 minutes. The protocol include a 3-minute rest period and a 6-minute stepping period.This measurement will be compared with those measured during a 6-minute walk test (gold standard for field tests) and a maximal cardiorespiratory exercise test on a cycloergometer (gold standard for laboratory tests)
Leg fatigue after 6MST measured by the modified Borg scale | 19 days
  The modified Borg scale is a numerical scale that allows individuals to subjectively rate their level of exertion during exercise. The scale ranges from 0 to 10, where 0 means "no exertion at all" and 10 means maximal exertion.
Maximum effort test after 6MST | 19 days
  The patient will perform the test on a cycloergometer and will be connected to a portable gas exchange analyzer via a face mask (Metamax 3B Cortex). After warming up, intensity will be increased by 10-15 W.min-1 until maximal effort is achieved, in line with recommendations. Participants will be asked to maintain a pedaling frequency of 60 ± 5 rpm. Blood pressure will be measured at rest, every 2 min during exercise and during 5 min of recovery.
Lower limb muscle power after 5STS test | 19 days
  A force platform (Multicomponent force plate, Kistler) will be positioned under the participant's feet. The muscular power developed by the lower limbs during the 5STS will be measured using this platform and the value will be compared with that calculated by the reference equation available in the literature.

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud CHAMBELLAN, MD, Principal Investigator — Hôpital Saint Philibert, GHICL
Locations (2):
- Centre de Pneumologie Institut universitaire de cardiologie et de pneumologie de Québec, Québec, Canada
- Hôpital Saint-Philibert (GHICL), Lomme, France

IPD SHARING:
Plan to Share IPD: No